CLINICAL TRIAL: NCT02282683
Title: Long-term Prednisone Use in Patients With Advanced Heart Failure (ACCF/AHA Stage D) and Hyperuricemia
Brief Title: Long-term Prednisone Use for End-stage Heart Failure
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Kun-shen Liu M.D., Professor, Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hebmu 201312
Record Dates: First submitted 2014-10-28; First posted 2014-11-04 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Heart Failure; Hyperuricemia
MeSH Terms: conditions — Heart Failure; Hyperuricemia | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisone (Experimental): Prednisone (10 to 20 mg/day, orally) combined with maximum tolerated guideline-directed medical therapy for at least 12 months.
  Interventions: Drug: prednisone
- Control (No Intervention): Maximum tolerated guideline-directed medical therapy

INTERVENTIONS:
Drug: prednisone — Prednisone (10 to 20 mg/day, orally) combined with maximum tolerated guideline-directed medical therapy for at least 12 months
  Arms: Prednisone

SUMMARY:
Patients with advanced (ACCF/AHA stage D) heart failure and hyperuricemia have high one-year mortality. Currently, there was no evidence-based therapy such as mechanically assisted circulatory support available in China. The investigators found glucocorticoid treatment such as prednisone could improve cardiac performance, potentiate renal responsiveness to diuretics in such patients. Therefore, it could be used as bridge therapy to help ACE inhibitors or beta blocker titration. With its help, most of the patients with stage D heart failure could be titrated to higher dose of ACE inhibitors and beta blockers during hospitalization. However, the efficacy of long-term, low-dose of prednisone use in such patients with limited life expectancy remain unclear. Therefore, the investigators designed this study to observe whether putting low-dose of prednisone on the patients with stage D heart failure for long term could further improve their survival. All patients will receive prednisone treatment during hospitalization and receive maximum tolerated guideline-directed medical therapy (GDMT). After discharge from hospital, the patients will be randomized to receive long-term, low-dose prednisone treatment or standard GDMT.

ELIGIBILITY:
Inclusion Criteria:

* Repeated (>2) hospitalizations or ED visits for HF in the past year
* Inability to exercise including exertion limited, exertion intolerance, resting symptoms or inotrope dependent
* Left ventricular ejection fraction ≤35%
* Serum uric acid level ≥500μmol/L
* Received prednisone treatment during hospitalization period and And more 5 of the followings

  1. Progressive deterioration in renal function (e.g., rise in BUN and creatinine)
  2. Weight loss without other cause (e.g., cardiac cachexia)
  3. Intolerance to ACE inhibitors due to hypotension and/or worsening renal function
  4. Intolerance to beta blockers due to worsening HF or hypotension
  5. Frequent systolic blood pressure <90 mm Hg
  6. Recent need to escalate diuretics to maintain volume status, often reaching daily furosemide equivalent dose >160 mg/d and/or use of supplemental thizide therapy
  7. Progressive decline in serum sodium, usually to <133 mEq/L
  8. Gastrointestinal symptoms (abdominal discomfort, nausea, poor appetite), disabling ascites, or severe lower-extremity edema

Exclusion Criteria:

* Any condition (other than heart failure) that could limit the use of prednisone
* Any concurrent disease that likely limits life expectancy;
* Active myocarditis, or an hypertrophic obstructive or restrictive cardiomyopathy;
* Myocardial infarction, stroke, unstable angina, or cardiac surgery within the previous 3 months;
* Indication for hemodialysis
* Uncontrolled systolic blood pressure > 160 mmHg
* Complex congenital heart disease
* Poorly controlled diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Mortality within 12 months | 12 months

SECONDARY OUTCOMES:
Event-free survival time (defined as time to first hospitalization due to heart failure deterioration or death) within 12 months | 12
Survival time (defined as time to death) within 12 months | 12 months
Change from baseline in serum uric acid | month 6 and month 12
Change from baseline in serum creatinine | month 6 and month 12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

REFERENCES:
- [Background] Liu C, Zhao Q, Zhen Y, Gao Y, Tian L, Wang L, Ji L, Liu G, Ji Z, Liu K. Prednisone in Uric Acid lowering in Symptomatic Heart Failure Patients With Hyperuricemia (PUSH-PATH) study. Can J Cardiol. 2013 Sep;29(9):1048-54. doi: 10.1016/j.cjca.2012.11.008. Epub 2013 Feb 6. PMID 23395281
- [Background] Liu C, Liu G, Zhou C, Ji Z, Zhen Y, Liu K. Potent diuretic effects of prednisone in heart failure patients with refractory diuretic resistance. Can J Cardiol. 2007 Sep;23(11):865-8. doi: 10.1016/s0828-282x(07)70840-1. PMID 17876376